CLINICAL TRIAL: NCT07282717
Title: Fibroblast Line Evaluation for COL5A eXpression and Thoracic Aortic Aneurysms: in Vitro Characterization of Cutaneous Fibroblasts in Adult Patients
Acronym: FLEX5 project
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Director, IRCCS Policlinico S. Donato
Other Study IDs: FLEX5 project
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-11

CONDITIONS: Mutations Affecting the COL5A Gene; Aneurysm Aortic
Keywords: COL5A; FIBROBLASTS; ascending and descending aortic aneurysms; thoracic aortic aneurysms
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adult patients with COL5A with TAAD: Adult patients (aged over 50 years) with COL5A mutation and aortic manifestations
- Adult patients with COL5A mutation without TAAD: Adult patients (aged over 50 years) with COL5A mutation in the absence of aortic manifestations
- Young patients with COL5A mutation and TAAD: Young patients (aged 18-50 years) with COL5A mutation and aortic manifestations
- Young patients with COL5A mutation without TAAD: Young patients (aged 18-50 years) with COL5A mutation in the absence of aortic manifestations

SUMMARY:
This study examines adults with COL5A gene mutations to understand why some develop aortic aneurysms while others do not. Participants provide a small skin biopsy, and researchers analyze fibroblasts to evaluate collagen production, extracellular matrix organization, and connective-tissue signaling pathways. The goal is to identify biological differences that may explain variable vascular risk and support future personalized monitoring and treatment strategies.

DETAILED DESCRIPTION:
Individuals with mutations in the collagent type V, alpha (COL5A) gene show variable clinical outcomes. While some develop aortic aneurysms, others with the same mutation remain free of cardiovascular complications. The mechanisms driving this variability are not fully understood.

This study aims to investigate biological differences at the cellular level by analyzing fibroblasts derived from a small skin biopsy. Fibroblasts play a key role in the production and organization of type V collagen and the extracellular matrix.

Researchers will:

Grow fibroblasts from participants' skin samples.

Assess cell growth, migration, and extracellular matrix formation.

Measure the quantity and type of collagen produced.

Evaluate molecules involved in collagen breakdown and repair.

The study compares individuals with COL5A mutations who have documented aortic aneurysms to those with the same mutation but no vascular involvement. Analyses will also consider differences among family members who share the same genetic variant.

By characterizing fibroblast behavior, the study seeks to clarify why some individuals develop aortic disease while others remain unaffected. Findings may help identify cellular features associated with increased or reduced vascular risk and guide future strategies for monitoring, prevention, and personalized care in patients with COL5A mutations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 and above
* Mutation in COL5A
* Signed informed consent

Exclusion Criteria:

* Corticosteroid or Steroids or Fluorochinolones treatment within six months before enrollment
* Subjects on chronic immunosuppressive therapies such as oral steroids, but also on chronic topical steroids in the area of investigation
* Subject on anticoagulant therapy
* History of coagulation factor defects/alterations (data found in anamnesis and medical records)
* A history of keloid formation (data found in anamnesis and medical records)
* Anesthetic drug allergy (data found in anamnesis and medical records)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Research hospital for rare cardiovascular diseases
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Fibroblasts phenotype | 24 months
  In vitro characterization and evaluation of fibroblasts phenotype in adult patients with COL5A mutations with or without aortic involvement (ascending and descending aortic aneurysms)
Differences molecular mechanisms in collagen | 24 months
  Identify differences in molecular mechanisms involved in collagen and ECM turnover pathways between family members according to the vascular manifestation and the genetic mutation in COL5A gene

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Genetic Centre IRCCS Policlinico San Donato, San Donato Milanese, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
IPD sharing will be defined at the active enrolment process of the study

REFERENCES:
- [Result] Phan QM, Fine GM, Salz L, Herrera GG, Wildman B, Driskell IM, Driskell RR. Lef1 expression in fibroblasts maintains developmental potential in adult skin to regenerate wounds. Elife. 2020 Sep 29;9:e60066. doi: 10.7554/eLife.60066. PMID 32990218
- [Result] Lu P, Takai K, Weaver VM, Werb Z. Extracellular matrix degradation and remodeling in development and disease. Cold Spring Harb Perspect Biol. 2011 Dec 1;3(12):a005058. doi: 10.1101/cshperspect.a005058. PMID 21917992
- [Result] Plikus MV, Wang X, Sinha S, Forte E, Thompson SM, Herzog EL, Driskell RR, Rosenthal N, Biernaskie J, Horsley V. Fibroblasts: Origins, definitions, and functions in health and disease. Cell. 2021 Jul 22;184(15):3852-3872. doi: 10.1016/j.cell.2021.06.024. PMID 34297930